CLINICAL TRIAL: NCT06041919
Title: A Phase 2 Study to Evaluate the Early Bactericidal Activity, Safety and Tolerability of Nebulised RESP301 in Adults With Newly Diagnosed, Rifampicin Susceptible Pulmonary Tuberculosis
Brief Title: Evaluating the Early Bactericidal Activity, Safety and Tolerability of Nebulised RESP301 in Adults With Tuberculosis
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Decision was made by the sponsor not to progress to Stage 2
Sponsor: Thirty Respiratory Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RESP30X-EBA
Record Dates: First submitted 2023-08-21; First posted 2023-09-18 (Actual); Results first posted 2025-07-15 (Actual); Last update posted 2025-07-15 (Actual); Status verified 2025-06

CONDITIONS: Rifampicin Susceptible Pulmonary Tuberculosis
Keywords: Early Bactericidal Activity (EBA)

STUDY DESIGN:
Intervention Model Description: Parallel control arm, randomised clinical study in two sequential stages, with no stratification
Who Masked: Outcomes Assessor
Masking Description: Microbiology staff will be blinded to treatment allocation.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- 1 (Active) (Experimental): Inhaled RESP301 6ml via nebulisation three times daily
  Interventions: Drug: RESP301
- 2 (Control) (Active Comparator): HRZE taken orally once daily
  Interventions: Drug: HRZE
- 3 (Active) (Experimental): Inhaled RESP301 6 ml via nebulisation once daily
  Interventions: Drug: RESP301
- 4 (Active) (Experimental): Inhaled RESP301 6 ml via nebulisation twice daily
  Interventions: Drug: RESP301
- 5 (Active) (Experimental): Inhaled RESP301 6 ml via nebulisation three times daily plus HRZE taken orally once dialy
  Interventions: Drug: RESP301; Drug: HRZE

INTERVENTIONS:
Drug: RESP301 — Nitric Oxide agent
  Arms: 1 (Active); 3 (Active); 4 (Active); 5 (Active)
Drug: HRZE — isoniazid 75 mg (H), rifampicin 150 mg (R), pyrazinamide 400 mg (Z), ethambutol 275 mg (E)
  Arms: 2 (Control); 5 (Active)

SUMMARY:
A Phase 2, Single-Centre, Open-Label, Parallel Control Arm, Randomised Clinical Study to Evaluate the Early Bactericidal Activity (EBA), Safety and Tolerability of Nebulised RESP301 in Adults with Newly Diagnosed, Rifampicin Susceptible Pulmonary Tuberculosis

DETAILED DESCRIPTION:
A total of approximately 15 participants will be recruited per treatment arm (total of approximately 75 participants in the study). Control arm participants will be split across sequential stages stages 1 and 2, with no stratification.

Stage 1: To determine the EBA of

* Treatment Arm 1 (Active; n = 15) - inhaled RESP301 6 ml dosed via nebulisation administered three times daily over 14 days
* Treatment Arm 2 (Control; n= 5) - HRZE taken orally once daily

On completion of Stage 1, recruitment will be paused and an interim analysis performed to determine whether the study should proceed to Stage 2.

Stage 2: To determine the EBA of

* Treatment Arm 2 (Control; n= 10) - HRZE taken orally once daily
* Treatment Arm 3 (Active; n = 15) - inhaled RESP301 6 ml dosed via nebulisation administered once daily over 14 days
* Treatment Arm 4 (Active; n = 15) - inhaled RESP301 6 ml dosed via nebulisation administered twice daily over 14 days
* Treatment Arm 5 (Active; n = 15) - inhaled RESP301 6 ml dosed via nebulisation administered three times daily in combination with HRZE taken orally once daily over 14 days

ELIGIBILITY:
Inclusion Criteria:

* Provide written, informed consent prior to all study-related procedures and agree to undergo all study procedures
* Body weight (in light clothing and with no shoes) between 40 and 90 kg, inclusive
* Newly diagnosed pulmonary TB
* Rifampicin susceptible pulmonary TB as determined by molecular testing
* Ability to produce an adequate volume of sputum as estimated from a pre-treatment overnight sputum collection sample (estimated 10 ml or more)
* Spirometry performed during screening with a FEV1 of ≥ 40%
* Be of non-childbearing potential or willing to use effective methods of contraception

Exclusion Criteria:

* HIV positive AND CD4 < 350 cells/mm3 OR are receiving antiviral therapy (ART)
* Methaemoglobin saturation (SpMet) >3%
* Female participant who is pregnant or breast-feeding
* Participants planning to conceive a child within the anticipated period of study participation and for at least 90 days after the last dose of IMP in the study
* Participation in other clinical studies with investigational agents within 8 weeks prior to screening
* Treatment received for this episode of TB with any drug active against M.tb
* Treatment with immunosuppressive medications such as TNF-alpha inhibitors within 2 weeks prior to screening, or systemic corticosteroids for more than 7 days within 2 weeks prior to screening.
* Treatment with nitric oxide and other nitric oxide donor agents, phosphodiesterase inhibitors and lung surfactant drugs, within 30 days prior to screening

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2023-09-27 (Actual); Primary Completion 2024-07-24 (Actual); Study Completion 2025-03-06 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- TASK Clinical Research Centre, Cape Town, Bellville, South Africa

IPD SHARING:
Plan to Share IPD: No
IPD is confidential until the CSR is published

RESULTS

PARTICIPANT FLOW:
Groups:
- 5 (Active): Inhaled RESP301 6 ml via nebulisation three times daily plus HRZE taken orally once daily
  RESP301: Nitric Oxide agent
  HRZE: isoniazid 75 mg (H), rifampicin 150 mg (R), pyrazinamide 400 mg (Z), ethambutol 275 mg (E)
Period: Overall Study
Arm/Group | 1 (Active) | 2 (Control) | 3 (Active) | 4 (Active) | 5 (Active)
Started | 15 | 5 | 0 | 0 | 0
Completed | 14 | 4 | 0 | 0 | 0
Not Completed | 1 | 1 | 0 | 0 | 0
Not completed — Lost to Follow-up | 1 | 0 | 0 | 0 | 0
Not completed — At the request of the investigator or the sponsor | 0 | 1 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: participants who received at least one dose of RESP301 or HRZE
Groups:
- Total: Total of all reporting groups
Arm/Group | 1 (Active) | 2 (Control) | 3 (Active) | 4 (Active) | 5 (Active) | Total
Number analyzed (Participants) | 15 | 5 | 0 | 0 | 0 | 20
Age, Continuous [Mean (Standard Deviation); unit: years] | 31.00 (10.09) | 31.20 (5.93) |  |  |  | 31.05 (9.08)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 1 |  |  |  | 3
  Male | 13 | 4 |  |  |  | 17
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 |  |  |  | 0
  Asian | 0 | 0 |  |  |  | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 |  |  |  | 0
  Black or African American | 15 | 5 |  |  |  | 20
  White | 0 | 0 |  |  |  | 0
  More than one race | 0 | 0 |  |  |  | 0
  Unknown or Not Reported | 0 | 0 |  |  |  | 0
Weight [Mean (Standard Deviation); unit: kg] | 53.05 (9.83) | 50.08 (6.76) |  |  |  | 52.31 (8.85)
Height [Mean (Standard Deviation); unit: m] | 1.69 (0.07) | 1.65 (0.05) |  |  |  | 1.68 (0.07)
BMI [Mean (Standard Deviation); unit: kg/m^2] | 18.70 (3.58) | 18.34 (1.70) |  |  |  | 18.61 (3.17)

OUTCOME MEASURES:

1. Primary Outcome: Early Bactericidal Activity (EBA) of Inhaled RESP301 Measured as Time to Positivity (TTP)
Description: Overnight sputum collection from which viable mycobacteria in the sample is quantified as TTP Observed EBA for 0-2, 0-7, 0-14, 0-15 and 14-15 days in TTP (hours) for treatment in each of the treatment groups
Time Frame: 0-2, 0-7, 0-14, 0-15 and 14-15 days
Population: Decision was made by the sponsor not to progress to Stage 2
Measure: Median (Inter-Quartile Range); unit: Hours
Arm/Group | 1 (Active) | 2 (Control) | 3 (Active) | 4 (Active) | 5 (Active)
Number analyzed (Participants) | 15 | 5 | 0 | 0 | 0
Hours
  0-2 | 3.5 [-5.2 to 5.6] | 63.5 [53.2 to 78.2] |  |  |
  0-7 | 2 [-6.9 to 15] | 140.2 [117 to 160] |  |  |
  0-14 | 2.5 [-7.8 to 9.1] | 167.8 [147.8 to 200.5] |  |  |
  0-15 | 6.2 [-8 to 16.1] | 225 [157.8 to 247.5] |  |  |
  14-15 | 7.5 [-3 to 17.5] | 2 [-5 to 47] |  |  |

2. Secondary Outcome: Early Bactericidal Activity (EBA) of Inhaled RESP301 Measured as Colony Forming Units (CFU)
Description: Overnight sputum collection from which viable mycobacteria in the sample is quantified as CFU Observed EBA for 0-2, 0-7, 0-14, 0-15 and 14-15 days in CFU (Log10 CFU/mL) for treatment in each of the treatment groups
Time Frame: 0-2, 0-7, 0-14, 0-15 and 14-15 days
Population: Decision was made by the sponsor not to progress to Stage 2
Measure: Median (Inter-Quartile Range); unit: Log10 CFU/mL
Arm/Group | 1 (Active) | 2 (Control) | 3 (Active) | 4 (Active) | 5 (Active)
Number analyzed (Participants) | 15 | 5 | 0 | 0 | 0
Log10 CFU/mL
  0-2 | 0.3 [-0.1 to 0.5] | -0.9 [-0.9 to -0.6] |  |  |
  0-7 | 0.2 [-0.2 to 0.4] | -1.2 [-1.6 to -0.8] |  |  |
  0-14 | 0.4 [-0.2 to 0.8] | -2.9 [-3.1 to -2.7] |  |  |
  0-15 | 0.3 [-0.4 to 0.7] | -2.4 [-3.6 to -1.4] |  |  |
  14-15 | 0 [-0.3 to 0.1] | 0.1 [0.1 to 0.1] |  |  |

3. Secondary Outcome: Safety and Tolerability of Inhaled RESP301 Measured as Number of Treatment Emergent Adverse Events (TEAEs)
Description: Incidence of Treatment Emergent Adverse Events (TEAEs) will be presented by severity, drug relatedness, seriousness, leading to early withdrawal and leading to death.
Time Frame: Stage 1: Dosing period 14 days + Follow-up period 14 days. Stage 2: Participants did not enter the treatment phase due to early study termination
Population: Decision was made by the sponsor not to progress to Stage 2
Measure: Number; unit: events
Arm/Group | 1 (Active) | 2 (Control) | 3 (Active) | 4 (Active) | 5 (Active)
Number analyzed (Participants) | 15 | 5 | 0 | 0 | 0
events
  Number of Grade 1 (Mild) TEAEs | 38 | 7 |  |  |
  Number of Grade 2 (Moderate) TEAEs | 13 | 2 |  |  |
  Number of Grade 3 (Severe) TEAEs | 2 | 0 |  |  |
  Number of Grade 4 (Life-threatening) TEAEs | 0 | 0 |  |  |
  Number of Unrelated TEAEs | 27 | 8 |  |  |
  Number of Related TEAEs | 26 | 1 |  |  |

ADVERSE EVENTS:
Time Frame: Stage 1: Dosing period 14 days + Follow-up period 14 days. Stage 2: Participants did not enter the treatment phase due to early study termination
Description: Stage 2 (Arm 3,4, and 5): Participants did not enter the treatment phase due to early study termination
Arm/Group | 1 (Active) | 2 (Control) | 3 (Active) | 4 (Active) | 5 (Active)
All-Cause Mortality (participants affected / at risk) | 0/15 | 0/5 | 0/0 | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/5 | 0/0 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 15/15 | 4/5 | 0/0 | 0/0 | 0/0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 1 (Active) (N=15) | 2 (Control) (N=5) | 3 (Active) (N=0) | 4 (Active) (N=0) | 5 (Active) (N=0)
Abdominal Pain (Gastrointestinal disorders) | 2 (2) | 1 (1) | NA | NA | NA
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0) | NA | NA | NA
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 0 (0) | NA | NA | NA
Gastritis (Gastrointestinal disorders) | 1 (1) | 0 (0) | NA | NA | NA
Post-Tussive Vomiting (Gastrointestinal disorders) | 1 (2) | 0 (0) | NA | NA | NA
Salivary Hypersecretion (Gastrointestinal disorders) | 1 (1) | 0 (0) | NA | NA | NA
Toothache (Gastrointestinal disorders) | 1 (1) | 0 (0) | NA | NA | NA
Gastroenteritis (Infections and infestations) | 1 (1) | 0 (0) | NA | NA | NA
Herpes Simplex (Infections and infestations) | 1 (1) | 0 (0) | NA | NA | NA
Vulvovaginal Candidiasis (Infections and infestations) | 1 (1) | 1 (1) | NA | NA | NA
Otitis Media (Infections and infestations) | 0 (0) | 1 (1) | NA | NA | NA
Urinary Tract Infection (Infections and infestations) | 0 (0) | 1 (1) | NA | NA | NA
Gamma-Glutamyltransferase Increased (Investigations) | 2 (3) | 0 (0) | NA | NA | NA
Weight Decreased (Investigations) | 1 (1) | 0 (0) | NA | NA | NA
Hyperkalaemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | NA | NA | NA
Back Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | NA | NA | NA
costcochondritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | NA | NA | NA
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | NA | NA | NA
Headache (Nervous system disorders) | 3 (3) | 1 (1) | NA | NA | NA
Insomnia (Nervous system disorders) | 1 (1) | 0 (0) | NA | NA | NA
Somnolence (Nervous system disorders) | 1 (1) | 0 (0) | NA | NA | NA
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 6 (6) | 0 (0) | NA | NA | NA
Chest Discomfort (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | NA | NA | NA
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | NA | NA | NA
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | NA | NA | NA
Cough (Respiratory, thoracic and mediastinal disorders) | 13 (17) | 0 (0) | NA | NA | NA
Pruritus (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1) | NA | NA | NA
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | NA | NA | NA

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2023-05-25): https://cdn.clinicaltrials.gov/large-docs/19/NCT06041919/Prot_000.pdf
  • Statistical Analysis Plan (2024-07-22): https://cdn.clinicaltrials.gov/large-docs/19/NCT06041919/SAP_001.pdf